CLINICAL TRIAL: NCT04242472
Title: SMS-based Mobile Health Intervention for Nutritional Status and Treatment Outcomes Among TB Patients in Addis Ababa, Ethiopia: A Cluster Randomized Trial (CRT)
Brief Title: SMS-based Mobile Health Intervention for Nutritional Status and Treatment Outcome Among TB Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Addis Ababa University (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Principal Investigator, Zekariyas Sahile, PhD candidate, Addis Ababa University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: TB-MeNu; D43TW009127 (NIH)
Record Dates: First submitted 2020-01-20; First posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Tuberculosis; Undernutrition
Keywords: Tuberculosis; Nutrition; Treatment outcome; SMS
MeSH Terms: conditions — Tuberculosis; Malnutrition

STUDY DESIGN:
Intervention Model Description: A Cluster Randomized Trial (CRT) with parallel design will be employed.
Who Masked: Outcomes Assessor
Masking Description: Participants and providers will not be blind to the study intervention. Nutrition and tuberculosis treatment outcomes will be assessed by two independent reviewers without knowledge of each participant's treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMS group (Experimental): Nutrition-related SMS messages in addition to standard of care TB treatment with directly observed therapy
  Interventions: Behavioral: SMS-based Mobile Health intervention
- Control group (No Intervention): Standard care of TB treatment with directly observed therapy alone

INTERVENTIONS:
Behavioral: SMS-based Mobile Health intervention — Nutritional related SMS text message mobile health intervention will be provided to Tuberculosis patients.
  Arms: SMS group

SUMMARY:
Ethiopia is one of the high burden Tuberculosis countries and Tuberculosis is still the leading cause of mortality due to communicable diseases in the country. Nutritional status is one of the predictors of TB treatment outcomes. Thus, the current practices need integration of nutritional intervention in the DOT using Mobile health intervention. However, to investigator's knowledge, there is no sufficient evidence on the effect SMS text Messaging Mobile Health intervention on nutritional status and TB treatment outcomes in Ethiopia.

DETAILED DESCRIPTION:
To ensure the quality of SMS intervention, nutritional related SMS text message will be developed systematically through reviewing literature, systematic reviews and guidelines and appropriate behavioral theories by involving experts and patients. Automated SMS will be sent from one computer database at the scheduled date and time. A validated questionnaire will be adapted and pre-tested to check for any error. Adequate sample size is calculated for both arms with the ratio of 1:1 allocation. Standardized Anthropometric measurement, FANTA Household Dietary Diversity Score and WHO TB treatment outcome classification will be used for assessing the outcome variables. The data collectors will be trained on the objective, screening of eligible participants, the procedure of data collection, and how to assure the quality and security of the data based on the protocol. Continuous supervision will be employed throughout the data collection and intervention period. The data will be collected electronically and will be exported to STATA for analysis. Intention to treat analysis and regression analysis model will be employed.

ELIGIBILITY:
Inclusion Criteria:

* Patient who is following their anti TB treatment for at most two weeks and below
* Patient who have their own mobile phone
* Patient who is able to read and understand national official language (Amharic)

Exclusion Criteria:

* Patient whose TB treatment regimen more than 6 months
* Patient who is pregnant and lactating mothers
* Patient who enrolled other Interventional research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2020-07 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Nutritional status change | Change from baseline BMI at end of 2 months and 6 months treatment
  The nutritional status of the patient will be assessed by Body Mass Index (BMI) that calculated through measuring the body weight and height of the patients using an electronic platform weight scale to the nearest 0.1 kg and height to the nearest centimeter using standardized meter.

SECONDARY OUTCOMES:
Dietary practice change | Change from baseline dietary practice at end of 6 months treatment
  Patient's dietary diversity practice will be assessed through a standardized tool adapted from FANTA Household Dietary Diversity Score
Treatment outcome | End of six months TB treatment
  Treatment outcomes will be classified as per WHO Tuberculosis treatment guideline. The classification is made based on the smear sputum examination result at second, five and end of six months treatment and/or treatment completion status.

CONTACTS AND LOCATIONS:
Overall Officials: Damen Haile Mariam, Study Chair — Addis Ababa University School of Public Health
Locations (1):
- Addis Ababa Health Bureau, Addis Ababa, Ethiopia

IPD SHARING:
Plan to Share IPD: No